CLINICAL TRIAL: NCT04970706
Title: Longitudinal Assessment of Cartilage Injury and Remodeling After Anterior Cruciate Ligament Rupture and Reconstruction: A Correlational Study of Functional Imaging and Biomarkers
Brief Title: Cartilage Injury and Remodeling After ACL Rupture and Reconstruction: Functional Imaging and Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: M2017401
Record Dates: First submitted 2021-06-27; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Volunteers were healthy people without ACL rupture
- Patients with ACL Rupture: All patients will undergo a standardized single-bundle technique with a hamstring or bone-patellar tendon-bone autograft.
  Interventions: Procedure: ACL reconstruction

INTERVENTIONS:
Procedure: ACL reconstruction — All patients will undergo a standardized single-bundle technique with a hamstring or bone-patellar tendon-bone autograft.
  Groups: Patients with ACL Rupture

SUMMARY:
The proposed study will establish novel relationships between intra-articular MSC recruitment, synovial inflammation, biomarkers of cartilage degeneration and joint inflammation, clinical patient factors, and downstream alterations in cartilage composition and morphology to provide novel insights into the pathoetiology of PTOA after ACL injury and reconstruction.

DETAILED DESCRIPTION:
In efforts to study the pathoetiology of post-traumatic osteoarthritis (PTOA), we propose a collaborative, prospective cohort study of 38 patients undergoing primary anterior cruciate ligament (ACL) reconstruction after ACL rupture. We will assess the longitudinal progression of patient-reported outcomes, knee laxity, MRI-based articular cartilage morphology and composition, and serum-borne biomarkers of cartilage degeneration up to 1 year of follow-up. Furthermore, stem cell mobilization, chemokine and pro-inflammatory cytokine concentrations, and inflammatory cell recruitment into synovial tissue will be measured from intraoperatively-collected samples. We will perform mixed multivariate linear regression modeling to elucidate potentially novel relationships between patient demographics, anatomy, biological factors, and downstream alterations in articular cartilage morphology and composition. We request $200,000 in funding over a two-year duration.

ELIGIBILITY:
Inclusion Criteria:

* - Males and females, aged 18 - 30 years
* Isolated, traumatic primary anterior cruciate ligament rupture requiring surgical reconstruction
* Surgical reconstruction performed using a single-bundle technique utilizing an autograft
* No history of ipsilateral traumatic knee injury or fracture
* No evidence of PCL injury or more than grade 1 injury to the MCL or LCL

Exclusion Criteria:

* - BMI < 18.5 or >35 kg/m2
* Injury occurred longer than 4 weeks before enrollment
* Intra-articular steroid injection within 3 months of injury
* Chondral defects greater than 3 cm2 or Outerbridge grade II or higher lesions

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The participating physicians at each site will identify potential subjects from their clinics' patients according to the inclusion/exclusion criteria listed below. Based on surgical volumes at both sites, patients generally undergo ACL reconstruction 8-12 weeks after initial screening. In the preoperative timeframe, all patients will undergo standard physical therapy to address pain, swelling, and motion deficits, as is standard of care at both institutions.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Objectives measure of knee stability | 3 months, 6 months, 12 months
  Knee stability (anterior-posterior laxity) will be measured utilizing the KT-2000 arthrometer, based on the side-to-side difference (SSD) observed between the injured and the healthy, contralateral knee. Subjects will be tested at 90 days, 180 days, and 1 year after surgery, with maximum manual force performed at 30 and 90 degrees of knee flexion.
COMP | 12 months after operation
  Cartilage Biomarker Analysis;
Interleukin-1 | 12 months after operation
  Chemokines and Pro-Inflammatory Cytokines in Synovial Fluid;
MMP-1 | 12 months after operation
  Soft Tissue Protease and Protease Inhibitor Analysis in Synovial Fluid
colony-forming units (CFU) | 12 months after operation
  The CFU assay is a common means of analyzing MSC concentration in bodily fluids
Cartilage morphology | 12 months after operation
  Quantitative MRI of cartilage morphology
Magnetic resonance imaging | 12 months after operation
  Quantitative MRI of Cartilage Composition

SECONDARY OUTCOMES:
Tegner Activity Scale | 12 months after operation
  knee evaluation are commonly used to document a patient's activity level
Lysholm Knee Scale | 12 months after operation
  knee evaluation are commonly used to document a patient's functional outcomes
International Knee Documentation Committee (IKDC) subjective Scale | 12 months after operation
  knee evaluation are commonly used to document a patient's functional outcomes

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Director — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided